CLINICAL TRIAL: NCT00076934
Title: A Phase I Study: Safety of RG2077 (CTLA4-IgG4m) in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: Safety of RG2077 in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Repligen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN006AI; NMS02 (Other: ITN)
Record Dates: First submitted 2004-02-06; First posted 2004-02-09 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: Ataxia; MRI; MS; CTLA4-IgG4m; Costimulatory Signals; Autoimmune Disorders
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Ataxia; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participants receive Regimen 1 for 4 months
  Interventions: Drug: RG2077 (CTLA4-IgG4m)
- 2 (Experimental): Participants receive Regimen 2 for 4 months
  Interventions: Drug: RG2077 (CTLA4-IgG4m)
- 3 (Experimental): Participants receive Regimen 3 for 4 months
  Interventions: Drug: RG2077 (CTLA4-IgG4m)
- 4 (Experimental): Participants receive Regimen 4 for 4 months
  Interventions: Drug: RG2077 (CTLA4-IgG4m)

INTERVENTIONS:
Drug: RG2077 (CTLA4-IgG4m) — RG2077

SUMMARY:
Multiple sclerosis (MS) is an autoimmune disorder. In this disease, the body's immune system attacks and destroys the cells that cover and protect nerves. This study will test the safety of a new drug called RG2077 that is designed to treat MS. The study will not determine whether RG2077 is effective in treating MS, only whether it is safe to use in patients with MS.

Study hypothesis: RG2077 will arrest MS if administered early in the course of MS and decrease accumulation of lesions on MRI.

DETAILED DESCRIPTION:
Effective treatment of autoimmune disorders is likely to arise not from improved immunosuppression, but from improved understanding of the normal mechanisms that generate and maintain self-tolerance. RG2077 may block a T cell costimulation pathway central to the pathophysiology of MS. A total of 20 patients with MS will be enrolled in this study. Each patient participates in the study for 4 months.

The dose-escalation portion of this study evaluated the safety of a single infusion of RG2077 (CTLA4-IgG4m) in 16 patients with MS and is now complete. Patients who participated in the single infusion portion of the study were assigned to one of four groups. Each group received a different dose of RG2077. The second portion of the study will evaluate the safety of 4 doses of RG2077 in 4 additional patients. In the multiple infusion portion of the study, all patients will receive the same dose of RG2077. Patients will be monitored for possible side effects of RG2077.

ELIGIBILITY:
Inclusion Criteria

* Confirmed diagnosis of MS, defined as an MRI consistent with MS plus two separate clinical events, or one clinical event and MRI consistent with demyelination plus a second MRI demonstrating new lesions
* Have declined all FDA approved therapies for MS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-01; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Safety assessment including a MRI, neurological and physical examinations | Throughout study

SECONDARY OUTCOMES:
Number of gadolinium (GD) enhancing lesions and T2 lesion volume on MRI | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Samia J. Khoury, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital/Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal.

REFERENCES:
- [Result] Viglietta V, Bourcier K, Buckle GJ, Healy B, Weiner HL, Hafler DA, Egorova S, Guttmann CR, Rusche JR, Khoury SJ. CTLA4Ig treatment in patients with multiple sclerosis: an open-label, phase 1 clinical trial. Neurology. 2008 Sep 16;71(12):917-24. doi: 10.1212/01.wnl.0000325915.00112.61. PMID 18794494
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY661 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY661 — ImmPort study identifier is SDY661
- Available data/document: Study protocol synopsis, -summary, -design, -adverse events, -medications,-demographics, - lab tests, -files: SDY661 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY661 — ImmPort study identifier is SDY661
- Available data/document: Individual Participant Data Set: ITN006AI/NMS02 — http://www.itntrialshare.org/project/Studies/ITN006AIPUBLIC/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available.
- Available data/document: Study protocol synopsis; -schedule of assessments; data and reports; adverse event(s); -specimens availability; -manuscripts and abstracts: ITN006AI/NMS02 — http://www.itntrialshare.org/project/Studies/ITN006AIPUBLIC/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available.